CLINICAL TRIAL: NCT01484470
Title: Umbilical Cord Transplantation for the Elderly Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Gamida Cell ltd (Industry)
Responsible Party: Principal Investigator, Patrick Stiff, Professor, Loyola University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202041
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Hematologic Malignancies
Keywords: Stem cell transplantation; Stem Cell expansion; Elderly
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unmanipulated arm (No Intervention): Participants that do not meet criteria for StemEx®, will be registered into the unmanipulated UCB arm and receive the standard conditioning regimen.
- Stemx Arm (Experimental): StemEx is a stem/progenitor cell-based product of ex-vivo expanded allogeneic UCB, which is administered to the subject in combination with the non-manipulated portion of the same cord blood unit (CBU). The CBU must be cryopreserved in two portions of which the larger (or equal) CBU portion contains at least 1.5 x 107 total nucleated cells (TNC)/Kg. This portion remains unmanipulated and is transplanted on Day 0. StemEx is derived from the smaller (or equal) CBU portion, which is expanded ex vivo for 21 days starting pre-transplant in the presence of cytokines TPO, IL-6, Flt-3L and SCF at a concentration of 50ng/ml and 5μM tetraethylenepentamine (TEPA)
  Interventions: Biological: StemEx

INTERVENTIONS:
Biological: StemEx — For patients allocated to StemEx® arm:
  * Day -20: Start small (or equal) portion expansion at processing site. (II) Conditioning Phase
  * Day -6 to -1: Subject receives a RIC regimen containing Fludarabine, Cyclophosphamide and Total Body Irradiation (TBI) (III) Transplantation and Follow-up Phase
  * Day 0: CBU unmanipulated portion transplantation (for StemEx® arm) or unmanipulated CBU transplantation.
  * Day 1: StemEx® transplantation.
  * Day 2 to 3 years: Post transplant follow-up.
  Arms: Stemx Arm

SUMMARY:
While cord blood transplants have been performed safely in elderly patients, many still relapse. The investigators propose to intensify the preparative regimen for this patient group in an attempt to decrease relapses, and combine this with an ex vivo expanded Umbilical Cord Blood (UCB) unit.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation is a life saving procedure in selected high-risk or recurrent hematologic malignancies and marrow failure syndromes. However its wide application is limited by availability of suitably HLA matched adult donors. Umbilical Cord Blood (UCB) has been increasingly used as an alternative hematopoietic stem cell source for these patients. To date, over 10,000 UCB transplants have been performed in both children32-38 and adults.35,39-44 Its advantages include easier procurement, decreased risk to donors, reduced risk of transmitting infections, the immediate availability of cryopreserved units, and acceptable HLA mismatches. The transplantation of UCB allows a greater degree of HLA mismatching without an unacceptably high incidence of graft versus host disease (GVHD). Adult patients receiving myeloablative cord blood transplants have a 90% chance of engraftment, but carry a 50% rate of transplant related mortality.

ELIGIBILITY:
Inclusion Criteria:

* Ages 55-73
* Patients will have one of the following malignancies:

  * Acute myelogenous leukemia (AML) deNovo in first CR with adverse cytogenetic abnormalities, M0, M6, M7 subtypes, extramedullary disease in remission or high CD34+ disease (> 50%)
  * AML in early relapse (5-10% blasts on bone marrow aspirate or biopsy), or beyond CR-1 with no circulating blasts
  * AML at any time if resulting from a previous myelodysplasia
  * Acute lymphocytic leukemia or lymphoblastic lymphoma (ALL) in first CR with adverse prognostic features: t (9; 22), extra medullary disease, or mature B cell phenotype
  * Acute lymphoid leukemia or lymphoblastic lymphoma in early relapse (5- 10% blasts on aspirate), or beyond CR-1
  * Acute Undifferentiated Leukemia or biphenotypic leukemia in CR1 or CR2
  * Transfusion dependent myelodysplastic syndrome (MDS) or refractory anemia with excess blasts (RAEB) or RAEB-in transition, CMMOL, or any myelodysplasia with 7q-, 5q-, 7-, 5- or resulting from prior anti cancer therapy.
  * Relapsed Non-Hodgkin's Lymphoma (NHL), including those that have relapsed after an autologous marrow/blood stem cell transplant
  * Chronic lymphocytic leukemia (CLL) patient who has had fludarabine and either failed or relapsed. Prior autologous transplant patients are eligible.
* Patients with adequate organ function and performance status criteria
* Subject must have at least one or the following back-up stem cell sources in case of engraftment failure:

  * Subject is willing to undergo BM harvest or peripheral blood progenitor cells (PBPC) collection for use in case of engraftment failure (when clinically applicable).
  * Subject has a second CBU as a possible back up.
  * Subject's haploidentical family member has been identified and agreed (by signing a written informed consent) to donate hematopoietic stem cells in case of engraftment failure.
* Evaluation by social service/psychologist
* Subject signs the written informed consent after being aware of the nature of the subject's disease and willingly consents to the treatment program after being informed of alternative treatments, potential risks, benefits and discomforts.
* Ability to understand and agree to compliance with strict evaluation, isolation,and medication schedules
* Designated primary care giver.
* Dental evaluation/treatment completed.
* ENT evaluation/treatment completed.
* All patient who survive to day 90 are eligible for measurement of T and B cell function and lymphocyte subset numbers to determine immune reconstitution post UCB transplantation with or without StemEx®

Exclusion Criteria:

* Patient with suitable related donor as defined per institutional guidelines
* Chemotherapy resistant or active AML, ALL, AUL, biphenotypic leukemia
* AML evolved from myelofibrosis
* MDS with 20% or greater bone marrow blasts at pre-transplant workup. Patients may receive therapy and if in remission, are eligible
* Prior allogeneic hematopoeitic stem cell transplant at any time
* Less than twenty-one days have elapsed since the subject's last radiation or chemotherapy prior to conditioning (except for hydroxyurea)
* Uncontrolled bacterial, fungal or viral infection at the time of study enrollment
* Seropositive or NAT positive for HIV, HTLV-1 and Hepatitis C
* Subjects with signs and symptoms of active central nervous system (CNS) disease
* Females who are pregnant or breastfeeding
* Allergy to bovine proteins or to aminoglycoside antibiotics (e.g. gentamicin) or to any product, which may interfere with the treatment.
* Patient unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up and research tests.
* Enrolled in another clinical trial or received an investigational treatment during the last 30 days, unless approved by the primary investigator.

Ages: 55 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Efficacy of StemEx | 100 days
  The primary endpoint is to demonstrate the efficacy of StemEx® vs. unmanipulated UCB transplantation in the elderly population (>55years of age) following RIC regimen by demonstrating engraftment with full donor chimerism (>98%) by Day 100 of more than 60% of the patients who received transplants expanded by the StemEx method.

SECONDARY OUTCOMES:
Time to engraftment | 42 days
  The day of neutrophil engraftment is defined as the first day of 3 consecutive days of an ANC greater than 500/microliter. The platelet recovery is the first of 3 consecutive measurements tested on different days of a platelet count greater than or equal to 20,000 without requiring platelet transfusions in the previous 7 days. Patients will be monitored for donor cell engraftment as evidenced by neutrophil recovery and donor chimerism in the marrow and/or peripheral blood at serial time points post transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stiff, MD, Principal Investigator — Loyola Universtiy Medical Center
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States